CLINICAL TRIAL: NCT01816802
Title: MERGE: MulticEnter ReGistry With Eeva
Brief Title: Registry Study of Traditional Morphology Grading Combined With Eeva in IVF Treatment
Acronym: MERGE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Progyny, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2012-AUX-009; TST 2193-p (Other: Auxogyn)
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Infertility
Keywords: In vitro fertilization; Assisted reproductive therapy; Time-lapse image recording; Image analysis software
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- In-vitro fertilization using Eeva: Patients undergoing in-vitro fertilization treatment who provide informed consent and use Eeva in their treatment cycle.
  Interventions: Device: In-vitro fertilization using Eeva

INTERVENTIONS:
Device: In-vitro fertilization using Eeva — Eeva will image embryos through cleavage stage (Day 3). Embryologists will use Eeva results along with traditional morphological grading to assist in selecting embryo(s) for transfer or freezing.

SUMMARY:
The purpose of this study is to record and evaluate the use of traditional morphology grading combined with Eeva in the treatment of in vitro fertilization.

DETAILED DESCRIPTION:
This is a prospective, observational, single-arm, nonrandomized, multicenter study. Data will be collected to establish eligibility, at baseline, during the stimulation and in vitro fertilization process, during embryo culture, at embryo transfer, at 12-18 days post egg retrieval to verify biochemical pregnancy, and then typically at 5-6 weeks gestational weeks to verify clinical pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing fresh in vitro fertilization treatment using their own eggs or donor eggs.

Exclusion Criteria:

* history of cancer.
* gestational carrier.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing in vitro fertilization treatment who provide informed consent and use Eeva in their treatment cycle.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate | 5-6 gestational weeks
  Determined by first pregnancy ultrasound outcome and optional 12-month phone follow-up

OTHER OUTCOMES:
Multiple Pregnancy Rate | 5-6 gestational weeks
  Determined by follow-up pregnancy ultrasound outcome
Spontaneous Miscarriage Rate | 5-6 gestational weeks
  Determined by follow-up pregnancy ultrasound outcome

CONTACTS AND LOCATIONS:
Overall Officials: Shehua Shen, MD, Study Director — Progyny, Inc.
Locations (12):
- United States (12):
  - HRC Fertility, Encino, California
  - Stanford Fertility and Reproductive Medicine Center, Palo Alto, California
  - Reproductive Partners, Redondo Beach, California
  - Pacific Fertility Center, San Francisco, California
  - Center for Advanced Reproductive Services (UCHC), Farmington, Connecticut
  - Fertility Centers of Illinois - River North, Chicago, Illinois
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Fertility Centers of Illinois, Highland Park IVF Center, Highland Park, Illinois
  - Long Island IVF, Melville, New York
  - University Hospital Fertility Center, Beachwood, Ohio
  - Institute for Reproductive Health, Cincinnati, Ohio
  - Fertility Center of San Antonio, San Antonio, Texas

REFERENCES:
- See also: Auxogyn, Inc. website — http://www.auxogyn.com